CLINICAL TRIAL: NCT02441725
Title: 1-minute Sit-to-stand Test: A Multicentre Validation Study of a Simple Exercise Capacity Test in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Validation of the 1-minute Sit-to-stand Test in Patients With COPD
Acronym: STAND-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STAND-UP Study
Record Dates: First submitted 2015-04-29; First posted 2015-05-12 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation Patients (Other): Validation of the 1-minute sit-to-stand test; for participants who consent including a extended daily assessment period of physical activity and patient-reported symptoms of exacerbations:
  Male and female COPD inpatients (≥40 years of age) from two pulmonary rehabilitation clinics (Klinik Barmelweid and Zürcher Höhenklinik Wald)
  Interventions: Other: 1-minute sit-to-stand test
- Acute Care Hospital Patients (Other): Validation of the 1-minute sit-to-stand test, including daily assessment of physical activity and patient-reported symptoms of exacerbations:
  Male and female COPD inpatients from two acute care hospitals (≥40 years of age; Stadtspital Waid and Spital Uster)
  Interventions: Other: 1-minute sit-to-stand test

INTERVENTIONS:
Other: 1-minute sit-to-stand test — Validation of the 1-minute sit-to-stand test in a COPD patient population

SUMMARY:
This is a study to provide an in-depth validation of the 1-minute sit-to-stand test as a measure of exercise capacity in patients with chronic obstructive pulmonary disease (COPD). Patients will perform the 1-minute sit-to-stand test and other validated exercise tests and questionnaires.

DETAILED DESCRIPTION:
Exercise capacity is a strong predictor for mortality, exacerbations and health-related quality of life (HRQL) in patients with chronic obstructive pulmonary disease (COPD). The 1-minute sit-to-stand test (1-min STS test) is a promising exercise capacity test that is simple to conduct and requires few resources.

This study will provide an in-depth validation of the 1-min STS test, specifically evaluating the tests reliability, validity, responsiveness to change and minimal clinically important difference. The study will also assess the predictive properties of the 1-min STS test with regards to detecting exacerbations, as well as identify patterns of physical activity and patient-reported symptoms of exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to GOLD criteria; post bronchodilator FEV1/FVC<70%
* Male and female patients ≥40 years of age
* Able to do at least 5 repetitions in the 1-min STS test at baseline assessment
* Written informed consent by the participant

Exclusion Criteria:

* Lower limb joint surgery in the preceding 3 months
* Too unstable medically to perform exercise tests
* Predominant neurological or musculoskeletal limitation to walking
* Cognitive reading impairment and/or difficulties managing the eDiary and step-counter

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
1-minute sit-to-stand test | Change from baseline after pulmonary rehabilitation programme
  Number of repetitions performed in the 1-minute sit-to-stand test

SECONDARY OUTCOMES:
5-repetition sit-to-stand test | Change from baseline after pulmonary rehabilitation programme
  Time taken to perform 5 sit-to-stand repetitions
6-minute walk test | Change from baseline after pulmonary rehabilitation programme
  Distance walked in 6 minutes
Quadriceps maximal voluntary contraction force | Change from baseline after pulmonary rehabilitation programme
Chronic Respiratory Questionnaire | Change from baseline after pulmonary rehabilitation programme
Hospital Anxiety and Depression Scale | Change from baseline after pulmonary rehabilitation programme
COPD Assessment Test | Change from Baseline after pulmonary rehabilitation programme
Baseline Dyspnoea & Transition Dyspnoea Index | Change from baseline after pulmonary rehabilitation programme
Feeling Thermometer | Change from baseline after pulmonary rehabilitation programme
Oxygen consumption (VO2) | Change from baseline (pre-exercise test) during and after test
Carbon dioxide production (VCO2) | Change from baseline (pre-exercise test) during and after test
Respiratory exchange ratio (RER) | Change from baseline (pre-exercise test) during and after test
Minute ventilation (VE) | Change from baseline (pre-exercise test) during and after test
Heart Rate | Change from baseline (pre-exercise test) during and after test
Blood oxygen saturation | Change from baseline (pre-exercise test) during and after test
Symptoms of exacerbations | Daily course over 3 months
  The EXAcerbations of Chronic Pulmonary Disease Tool (EXACT)
Physical activity | Daily course over 3 months
  As measured by a pedometer
Localisation | Daily course over 3 months
  As measured by GPS information

CONTACTS AND LOCATIONS:
Overall Officials: Anja Frei, pHd, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland